CLINICAL TRIAL: NCT02575183
Title: Varenicline (Chantix) Treatment for Waterpipe Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WI195422
Record Dates: First submitted 2015-03-25; First posted 2015-10-14 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2020-09

CONDITIONS: Nicotine Dependence
Keywords: Waterpipe smoking; Nicotine dependence; Smoking cessation; Varinecline, Chantix therapy; Behavioral therapy
MeSH Terms: conditions — Tobacco Use Disorder; Water Pipe Smoking; Smoking Cessation | interventions — Varenicline; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Chantix) (Experimental): 76 participants will be assigned to 4 behavioral therapy cessation for smoking cessation and will be randomized to receive Varinecline with instructions for administration for 12 weeks starting 1 week before "Smoking Quit Date" as suggested by the manufacturer: Days 1 to 3: 0.5 mg orally once a day Days 4 to 7: 0.5 mg orally twice a day Days 8 to end of treatment: 1 mg orally twice a day. Intervention 'Varinecline (Chantix)' and Intervention 'Behavioral Therapy'
  Interventions: Drug: Varinecline (Chantix); Behavioral: Behavioral Therapy
- Placebo (Placebo Comparator): 76 participants will be assigned to 4 behavioral therapy cessation for smoking cessation and will be randomized to receive a Placebo for Varinecline with instructions for administration for 12 weeks starting 1 week before "Smoking Quit Date" as suggested by the manufacturer: Days 1 to 3: a placebo (matched to 0.5 mg of Varenicline) orally once a day Days 4 to 7: a placebo (matched to 0.5 mg of Varenicline) orally twice a day Days 8 to end of treatment: a placebo (matched to 1 mg of Varenicline) orally twice a day.
  Intervention 'Placebo (for Varenicline)' and Intervention 'Behavioral Therapy'
  Interventions: Drug: Placebo (for Varenicline); Behavioral: Behavioral Therapy

INTERVENTIONS:
Drug: Varinecline (Chantix) — A randomized double-blind placebo-controlled trial that will evaluate the effect of Varenicline (Chantix), in 2 parallel groups of habitual waterpipe smokers who are willing to quit (n=152). 76 subjects will be randomized to receive varenicline (Chantix). The participants, study investigators and personnel who will be interviewing the participants and collecting the clinical data, will be blinded to the assigned treatment.
  Arms: Varenicline (Chantix)
Drug: Placebo (for Varenicline) — A randomized double-blind placebo-controlled trial that will evaluate the effect of Varenicline (Chantix), in 2 parallel groups of habitual waterpipe smokers who are willing to quit (n=152). 76 subjects will be randomized to receive a varenicline-matched. The participants, study investigators and personnel who will be interviewing the participants and collecting the clinical data, will be blinded to the assigned treatment.
  Arms: Placebo
Behavioral: Behavioral Therapy — This intervention is for all study participants and it involves 4 visits to the hospital. Each visit include a 30-min one-on-one individual session with the specialized therapist during which participants will be taught how to manage any withdrawal symptoms they experience, how to anticipate high-risk situations, deal with smoking triggers, achieve and maintain their goal to stop waterpipe smoking.

SUMMARY:
The lack of proven waterpipe smoking cessation interventions makes it important to explore interventions proven effective for cigarette smoking cessation. The investigators hypothesize that Varenicline (Chantix) administrated for 12 weeks is associated with higher sustained quit rate at 12 weeks compared to placebo. The investigators propose to conduct a randomized double-blind placebo-controlled trial that will evaluate the effect of Varenicline (Chantix), in two parallel groups each consisting of 76 habitual waterpipe smokers who are willing to quit. Potential participants will be approached in cafés, word-of-mouth and through media and will be invited to the American University of Beirut Medical Center to complete study procedures. Both study groups will receive the same behavioural intervention in combination with either Varenicline (Chantix), an FDA approved drug indicated for use as an aid to smoking cessation treatment, or placebo. Participants will complete study procedures in four visits. During visit-1 the informed consent process, baseline assessments and randomization will be completed and Varenicline (Chantix) or Placebo will be initiated together with the behavioural interventions. The behavioural intervention will be continued over the next 2 visits. An end of treatment visit 12 weeks after quit date will be dedicated to assessing sustained quit rate and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Daily waterpipe smokers from the community of Beirut,
* aged 18 years or older
* willing to quit

Exclusion Criteria:

* Cigarette and/or cigars smokers,
* active malignancy
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Prolonged abstinence from waterpipe smoking at three months post-cessation | up to 3 months
  Percent of participants who achieved sustained abstinence after a two-weeks grace period from quit date until final follow-up. This outcome will be assessed by self-reports and measured exhaled Carbon Monoxide and urine cotinine levels.

SECONDARY OUTCOMES:
Continuous abstinence prevalence | up to 3 months
  Percent of participants who achieved sustained abstinence since quit date until the final follow-up. This outcome will be assessed by self-reports and measured exhaled Carbon Monoxide and urine cotinine levels.
Seven-day point prevalence abstinence | Last 7 days before final visit
  Percent of subjects who had no waterpipe use during the seven-day preceding final follow-up. Outcome will be assessed by self-reports, exhaled Carbon Monoxide and urine cotinine levels.
Participants' adherence rate to the study procedures | up to 3 months
  Measured by the number of pills used and the number of behavioural therapy sessions attended.
Change in weight | Baseline and 3 months
  Change in weight between enrolment (visit-1) and end of treatment (visit-4, 3 month after quit date).
Change in blood pressure | Baseline and 3 months
  Change in blood pressure between enrolment (visit-1) and end of treatment (visit-4, 3 month after quit date).
Evaluation of the Behavioral intervention | Up to 3 months
  Participant's perception of the appropriateness and usefulness of the acquired behavioral interventions assessed using a questionnaire at the end of treatment
Severity of symptoms | Every two weeks, up to 3 months
  severity of abstinence symptoms and/or side effects related to Varenicline (Chantix) measured using the Minnesota Nicotine Withdrawal Scale and Varenicline (Chantix) side effects questionnaire during each follow-up phone call and at visits 2, 3 and 4.
Change in anxiety scores | Baseline and 3 months
  measured by the "Hopkins Symptoms Checklist-25 (HSCL-25)"between enrollment (visit-1, 1 week before quit date) and end of treatment (visit-4).
Change in depression scores | Baseline and 3 months
  measured by the "Hopkins Symptoms Checklist-25 (HSCL-25)"between enrollment (visit-1, 1 week before quit date) and end of treatment (visit-4).

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon